CLINICAL TRIAL: NCT04937400
Title: Delirium in Children Undergoing Stem Cell Transplantation: Epidemiology and Outcomes
Brief Title: Delirium in Children Undergoing Stem Cell Transplantation
Status: Active, not recruiting | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 20-08022572; R01CA244500 (NIH)
Record Dates: First submitted 2021-06-22; First posted 2021-06-24 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Stem Cell Transplant Complications; Delirium
Keywords: pediatric; stem cell transplant; outcomes; epidemiology
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric Stem Cell Transplant Patients: A consecutive cohort of children admitted to the hospital for stem cell transplantation
  Interventions: Other: Daily screening for delirium

INTERVENTIONS:
Other: Daily screening for delirium — Each child will be screened twice daily for delirium throughout the transplant hospitalization
  Other Names: Cornell Assessment for Pediatric Delirium

SUMMARY:
Children undergoing stem cell transplants are at risk for delirium, a temporary change in thinking and behavior. This study will define delirium rates, risk factors, and outcomes. Our eventual goal is to reduce delirium in this population.

DETAILED DESCRIPTION:
Delirium -- defined as an acute change in awareness and cognition that occurs in the setting of an underlying illness -- is a common complication of hematopoietic stem cell transplantation (HSCT) in adults, with associated morbidity and mortality. This has never been studied in children, where risk factors may vary substantially from adults. The objectives of this study are: to define the epidemiology of delirium, and measure its effect on outcomes.

This prospective longitudinal cohort study will prospectively establish the incidence of delirium in 1000 children in the peri-transplant period, and identify modifiable risk factors that predispose to delirium development. This study will also define the effect of delirium on important clinical outcomes, including neurocognitive function. This study will be executed by a research consortium of five leading pediatric oncologic transplant centers in North America, in collaboration with the leading pediatric delirium research group in the United States.

This innovative proposal will leverage the combined experience of the pediatric delirium and HSCT teams to expand urgently needed delirium research into a unique and unstudied population. By reducing delirium rates, outcomes after pediatric HSCT can be optimized.

ELIGIBILITY:
Inclusion Criteria:

* Age 0-21 years old
* Admitted for purpose of stem cell transplant

Exclusion Criteria:

* Age >21 years old
* Admitted for reason other than stem cell transplant (example: late post-transplant complications).

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subjects will include all patients admitted to the five participating pediatric stem cell transplant sites for the purpose of HSCT during the study period. Enrollment goal is 1000 subjects overall, and 240 subjects for neurocognitive testing. Subjects will be seriously ill. Every patient admitted for HSCT will be eligible for inclusion, unless they are >21 years old. Subjects will be enrolled regardless of gender, race, or ethnicity. No subgroups will be excluded, as delirium likely affects children of all ages and developmental trajectories, with no predilection based on gender, race, or ethnicity.
Sampling Method: Probability Sample
Enrollment: 1040 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Delirium incidence | 1-50 days
  Number of patients who develop delirium during the course of their transplant hospitalization

SECONDARY OUTCOMES:
Hospital length of stay | 1-365 days
  Length of transplant hospitalization will be measured in days.
Mortality rate | 1-5 years
  Count will include number of patients with either in-hospital or post-discharge mortality.
Readmission rate | 1-365 days
  Count will include number of patients who are readmitted to the hospital within 30-days of discharge.
Change in neurocognitive functioning as measured by the NIH Toolbox Cognition Battery | pre-transplant, 3 months after transplant, 12 months after transplant
  Neurocognitive functioning will be measured by the NIH Toolbox Cognition Battery, and reported as a total composite score ranging from 50-150. An average score, adjusted for age, is 100. A score lower than 100 indicates lower cognitive functioning than average; a score higher than 100 indicates higher cognitive functioning than average.

CONTACTS AND LOCATIONS:
Overall Officials: Chani Traube, Principal Investigator — Weill Medical College of Cornell University
Locations (6):
- United States (5):
  - University of California San Francisco, San Francisco, California
  - Dana Farber Cancer Center, Boston, Massachusetts
  - Weill Cornell Medical College, New York, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St Jude Children's Research Hospital, Memphis, Tennessee
- Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be shared via NIH-approved repositories within 12 months after publication of primary results. The sharing of unpublished information may be subject to confidentiality issues and will need to be discussed with the appropriate institutions before any request is granted. Access will be granted to qualified researchers with a methodologically sound proposal and appropriate agreements, for academic research, meta-analyses, and other approved studies.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: De-identified IPD will be available no later than 12 months after publication of the primary results and for at least 5 years thereafter.
Access Criteria: Access will be granted to qualified researchers with a methodologically sound proposal. Researchers must agree to a data use agreement, and requests will be reviewed by the study team and the Data Coordinating Center.

REFERENCES:
- [Background] Traube C, Gerber LM, Mauer EA, Small K, Broglie L, Chopra YR, Duncan CN, Ebens CL, Fitzgerald JC, Freedman JL, Hudspeth MP, Hurley C, Mahadeo KM, McArthur J, Shapiro MC, Sharron MP, Wall DA, Zinter MS, Greenwald BM, Silver G, Boulad F. Delirium in Children Undergoing Hematopoietic Cell Transplantation: A Multi-Institutional Point Prevalence Study. Front Oncol. 2021 Apr 22;11:627726. doi: 10.3389/fonc.2021.627726. eCollection 2021. PMID 33968727